CLINICAL TRIAL: NCT03472222
Title: Arsha Vidya Program for Preventing Drug Abuse Among Disadvantaged Children in Urban Slums
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NMP Medical Research Institute (Other)
Collaborators: Arsha Vidya Study Centre (Unknown); United Research International (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: NMP/10122
Record Dates: First submitted 2018-02-24; First posted 2018-03-21 (Actual); Last update posted 2019-05-24 (Actual); Status verified 2019-01

CONDITIONS: Drug Abuse
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: Quasi experimental design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arsha Vidya Program (Experimental): Arsha Vidya outreach community program was conducted with children. An unique well-planned teaching program developed to educate Indian cultural values & heritage to young children and adults with yoga, chants, religious and spiritual practices through stories, group activities and plays.
  Interventions: Behavioral: Arsha Vidya program

INTERVENTIONS:
Behavioral: Arsha Vidya program — Integrated intervention program includes counselling and supportive care with the support of Arsha Vidya program

SUMMARY:
Substance abuse remain critical problems in both developed and developing countries. Under privileged communities where health and economic system is weakest, use of drugs and illicit substances starts during adolescence and young adulthood. This not just affect physical development, mental health and social integration, but also family formation and stability, deviant behaviour, sexual behaviour and involvement, educational pursuits, livelihood pursuits. Therefore, emphasises the need for preventive education at this impressionable age.

ELIGIBILITY:
Inclusion Criteria:

* Parental consent to participate

Exclusion Criteria:

* Family not involved in de-addiction program
* Planning to move the area
* Mental incapacity to consent or participate

Ages: 7 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2018-02-21 (Actual); Primary Completion 2018-08-30 (Actual); Study Completion 2018-09-06 (Actual)

PRIMARY OUTCOMES:
Percent days abstinent of tobacco, alcohol and drugs | change from baseline to 12-weeks
  Daily Dairy was given to assess days abstinent of tobacco, alcohol and drugs

SECONDARY OUTCOMES:
Well being | change from baseline to 12-weeks
  The Well-Being Index (WBI), 5-item scale used to assess changes in general well-being.

OTHER OUTCOMES:
Craving | change from baseline to 12-weeks
  Frequency, intensity and duration of craving assessed visual analogue Scale

CONTACTS AND LOCATIONS:
Overall Officials: Buddhatmananda Saraswati, Study Chair — Arsha Vidya Study Centre, India; Rajubhai P Odedra, Principal Investigator — NMP Medical Research Institute; Divya Gaur, Study Director — United Research International
Locations (1):
- NMP Medical Reserach Institute, Ahmedabad, Gujarat, India

IPD SHARING:
Plan to Share IPD: Undecided